# Urinary Tract Dilations in Prenatal and Postnatal Life

ID: 0292/21/2023-00590

Dr. Svetlana Jánošová, PhD.

19.12.2023

# Information for the patient and an informed consent form with mandatory patient instruction, or his legal representative

## Dear patient

Ask for consent to participate in the study that we want to implement in medical facilities: SonoClinic s.r.o., Emporia, s.r.o. and NefroSa s.r.o. In the study, we will work with the data obtained during the ultrasound examination of your fetus and, in indicated cases, also of your child after birth, which we will send to the nephrology clinic Nefrosa s.r.o. The data will be processed anonymously and will be used only for research purposes in order to improve the management of patients with dilative urinary tract disease. We also ask for the addition of some data that we will need in the analysis of the obtained data. Thank you in advance for your cooperation.

### **Study title:**

Urinary Tract Dilations in Prenatal and Postnatal Life

### Important data:

| Name and surname |
|------------------------------------------------------|
| Method of pregnancy |
| Occurrence of kidney anomalies in you, the father |
| and siblings of the fetus |
| Surname. name of the child after birth (only for the |
| purpose of finding the child at the nephrologist) |
| Phone contact |
| Mail address |

| agree to participate in the study and I also agree to the processing of personal data. |
|---|
| Signature of the patient |